CLINICAL TRIAL: NCT06087575
Title: Early Feasibility Study of the Supira System in Patients Undergoing High-Risk Percutaneous Coronary Intervention (HRPCI) - The SUPPORT I Trial
Brief Title: Early Feasibility Study of the Supira System in Patients Undergoing HRPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supira Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-10003
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; High-risk Percutaneous Coronary Intervention; Interventional Cardiology
Keywords: left ventricular assist device (LVAD); peripheral mechanical circulatory support (MCS); Supira System
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The study is a prospective, non-randomized, single-arm, multicenter, feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Supira System (Experimental): Ventricular support indicated for use during elective or urgent high-risk percutaneous coronary interventions.
  Interventions: Device: Supira System

INTERVENTIONS:
Device: Supira System — The Supira System is a minimally invasive, miniaturized percutaneous ventricular assist device (pVAD) system that is intended to provide temporary (≤4 hours) hemodynamic support to patients undergoing a HRPCI procedure. The Catheter is inserted percutaneously via the femoral artery, across the aortic valve, and into the left ventricle under fluoroscopic guidance, with a portion remaining in the ascending aorta. The left ventricle is unloaded by pumping blood from the ventricle into the ascending aorta and systemic circulation.

SUMMARY:
The objective of this study is to assess the feasibility and safety of the Supira System in providing temporary cardiovascular hemodynamic support in patients undergoing HRPCI. The clinical data may be used to support subsequent regulatory applications and further evaluation of the Supira System.

DETAILED DESCRIPTION:
The Supira System is a temporary (≤ 4 hours) ventricular support device indicated for use during elective or urgent HRPCI performed in hemodynamically stable patients with severe coronary artery disease when a heart team, including a cardiac surgeon, has determined HRPCI is the appropriate therapeutic option.

ELIGIBILITY:
Subjects will be eligible for inclusion in this study if all of the following criteria apply:

1. Age ≥18 and ≤90 years
2. Subject is hemodynamically stable and will undergo elective or urgent (not emergent) HRPCI, where hemodynamic support is needed, as determined by the institutional heart team
3. Informed consent granted by the patient or legally authorized representative

Subjects who meet any one of the following criteria will be excluded from study participation:

1. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure

   a. Note: Cardiogenic shock is defined as: systemic hypotension (systolic blood pressure (BP) <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90 mmHg) plus one of the following: any requirement for inotropes/pressors prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion or use of intra-aortic balloon pump (IABP), or any other circulatory support device.
2. Stroke within 6 months of the index procedure, or any prior stroke with permanent neurologic deficit
3. Evidence of left ventricular thrombus as assessed by Transthoracic Echocardiogram (TTE)
4. Aortic valvular disease or regurgitation categorized as moderate or greater (≥2+ on a 4-grade scale as assessed on TTE)
5. Aortic stenosis categorized as moderate or greater (gradient >20 mmHg or valve area <1.5 cm^2 as assessed on TTE)
6. Previous aortic valve replacement or reconstruction
7. Ascending or descending aortic dissection or aortic aneurysm >4.5 cm
8. Aortic and iliofemoral anatomical conditions that preclude safe delivery and placement of the investigational device
9. Presence of decompensated liver disease; severe liver dysfunction (Child class C)
10. Ongoing renal replacement therapy with dialysis
11. Infection of the proposed procedural access site or systemic active infection requiring ongoing antibiotic therapy
12. Heparin-induced thrombocytopenia, current or any prior occurrences
13. Known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or known hypersensitivity to heparin, aspirin, adenosine diphosphate (ADP) receptor inhibitors, or nitinol
14. Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000/mm³ or spontaneous International Normalized Ratio (INR) ≥1.5 or known fibrinogen ≤1.5 g/L)
15. Any condition or scheduled surgery that will require discontinuation of antiplatelet and/or anticoagulant therapy within 90 days of the index procedure
16. Planned coronary intervention within 30 days post index procedure
17. Breastfeeding or pregnant
18. Currently participating in active follow-up phase of another clinical study of an investigational drug or device
19. Active COVID-related infection or prior COVID-19 diagnosis with sequelae that could confound endpoint assessments
20. Other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to provide written informed consent and/or to comply with study procedures
21. Considered to be part of a vulnerable population (defined as individuals with mental disability, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent; vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Feasibility: Successful initiation and maintenance of hemodynamic support | From device delivery through removal (up to 4 hours)
  Successful initiation and maintenance of hemodynamic support without severe hypotension throughout the index procedure. Sustained hypotension is defined as sustained mean arterial pressure (MAP) < 60 mmHg requiring inotropic/pressor medications or alternative mechanical circulatory support.
Safety: Rate of composite major device-related adverse events (MDRAEs), from device insertion through device removal (inclusive of Supira procedure-related SAEs). | From device delivery through device removal (up to 4 hours)
  MDRAEs are defined as any serious adverse events that are adjudicated by the Clinical Events Committee (CEC) as definitely or probably related to the Supira System.

SECONDARY OUTCOMES:
Technical Success | From device delivery through device removal (up to 4 hours)
  Rate of technical success, defined as completion of the entire Supira System procedure, including delivery, operation without device malfunction, and successful removal of the Catheter
Procedural Success | From device delivery through device removal (up to 4 hours)
  Rate of procedural success, defined as the rate of technical success without procedural SAEs.
Rate of composite MDRAEs from device removal through hospital discharge or 72 hours post-procedure, whichever occurs first. | From device removal through hospital discharge or 72 hours post-procedure (whichever occurs first) through 30 days post device removal.
Rate of composite MDRAEs from hospital discharge or 72 hours post-procedure (whichever occurs first) through 30 days post device removal. | From hospital discharge or 72 hours post-procedure (whichever occurs first) through 30 days post device removal.
Rate of composite MDRAEs from 30 days to 90 days post device removal. | From 30 days to 90 days post device removal.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California Davis (UC Davis) Medical Center, Sacramento, California
  - Piedmont Heart Institute Cardiovascular Research, Atlanta, Georgia
  - Mount Sinai, New York, New York
  - Montefiore Medical Center Cardiology Research, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No